CLINICAL TRIAL: NCT04021797
Title: Autonomic Mechanisms of Sleep-dependent Memory Consolidation
Acronym: MemS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to COVID-19
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Memory+Stimulation; A127552 (Other Grant/Funding Number: National Center for Advancing Translational Science)
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Memory; Sleep

STUDY DESIGN:
Intervention Model Description: We will employ a within-subjects, crossover, sham-controlled design. Each participant will be exposed to both active and sham conditions over two visits (5-days apart).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant's will not be aware which configuration represents the sham vs active stimulation condition. Data analyses will be conducted blind to sham or active stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Sham (Sham Comparator): For the sham condition, the electrodes will be attached to an ear location that has not been shown to engage the vagus nerve. The stimulation frequency, intensity and duration will be aligned with the same parameters presented for the active tVNS condition (8Hz frequency, 5.0 mA electrical current and 200 ms pulse width).
  Interventions: Device: transcutaneous vagal nerve stimulation
- Active (Experimental): For the active condition, the electrodes will be attached to the ear at a place previously demonstrated to stimulate the vagus nerve. The stimulation frequency, intensity and duration will be aligned with the same parameters presented for the sham condition (8Hz frequency, 5.0 mA electrical current and 200 ms pulse width).
  Interventions: Device: transcutaneous vagal nerve stimulation

INTERVENTIONS:
Device: transcutaneous vagal nerve stimulation — The transcutaneous stimulator engages the cymba conchae in the left inner ear, compared to the left earlobe in the sham stimulation condition.

SUMMARY:
The goal of the proposed project is to identify the impact vagal activity during sleep for memory formation. Nearly 100 years of research contends that sleep plays a critical role in memory consolidation (i.e. the transformation of recent experiences into stable, long-term memories), yet much of this literature has focused on the central nervous system and technologies like electroencephalography (EEG) to unpack neural correlates involved in memory processing. Sleep is also a unique period of autonomic variation and an expansive literature has indicated the critical importance of the autonomic nervous system for memory formation. This project would be amongst the first to examine the autonomic nervous system during sleep as a critical, causal pathway linking sleep to memory processing. The investigators will assess the impact of non-invasive, transcutaneous vagal nerve stimulation on sleep and post-sleep memory performance. Autonomic physiology, including electrocardiography and impedance cardiography, will be gathered at baseline, before the memory task and continuously during sleep to examine vagal tone (i.e. heart rate variability) and sympathetic activation (i.e. pre-ejection period) in response to both active and sham stimulation conditions. Polysomnography will also be gathered during the nap to examine sleep architecture. The proposed research will address a critical gap in the literature by: 1) examining the causal role of the ANS for memory functioning in humans, 2) extending the current understanding of sleep's impact on memory processing, and 3) set the groundwork for novel, sleep-based interventions with the goal of improving cognitive health.

DETAILED DESCRIPTION:
Poor sleep is associated with significant cognitive health decline. Recently, sleep disturbances have emerged as notable predictive and exacerbating factors in the onset and development of neurodegenerative disease. Decades of research have implicated that sleep plays a critical role in memory consolidation (i.e. the transformation of recent experiences into stable, long-term memories), the decline of which is critical in the early stages of dementia. This literature affords that sleep, a period of reduced external interference, provides an optimal window for memory consolidation and that electrophysiological features that emerge during sleep are integrally involved in the consolidation process. Most of this literature has focused on the central nervous system and technologies like electroencephalography (EEG) to unpack neural correlates involved in memory processing. However, little impact from this work has translated into practical treatments and recent reviews of the literature question these sleep - memory associations. This lack of clarity suggests that there may be other factors critical to our understanding of sleep-dependent memory consolidation that have not been given due consideration. This proposal suggests that the autonomic nervous system (ANS) during sleep may reflect a critical, though understudied, pathway linking sleep and memory.

An expansive body of research has supported the role of the ANS for memory formation. Rodent studies have found that the storage of new information in memory is either enriched or impaired following learning acquisition by directly modifying peripheral activity through the vagus nerve. The vagus nerve is responsible for communicating information about peripheral excitation and arousal via projections to the brainstem, which then projects to memory-related areas including the amygdala complex, hippocampus, and prefrontal cortex. Indeed, in humans, researchers have demonstrated that direct stimulation of the vagus nerve, via surgical implants, can enhance declarative memory in epileptic patients and in patients with Alzheimer's Disease. Recently, in a sample of healthy older adults, non-invasive (transcutaneous) vagal nerve stimulation during wake boosted memory for face-name associations. Importantly, previous research has demonstrated the predominance of parasympathetic/vagal activity during sleep, particularly during slow wave sleep, which has received critical attention for its causal role in declarative memory consolidation. More so, the PI's work has shown that sleep acts as a regulatory influence over vagal activity and that vagally-mediated activity during sleep can predict post-sleep memory improvement. Yet, few investigations have examined the causal impact of vagal activity during sleep for memory outcomes, which is the central aim of this application.

In this project, the investigators will utilize a within-subject, sham-controlled, counterbalanced design to determine the impact of active (inside of left ear) vs. sham (left earlobe) transcutaneous vagal nerve stimulation (tVNS) on: 1) sleep architecture, 2) autonomic activity during sleep, and 3) memory performance post-sleep. To this end, the investigators will utilize a daytime nap protocol, a common methodological tool used to assess the role of sleep for cognition. A nap approach allows for strict circadian-control of cognition and provides for an examination of tVNS's impact on a full cycle of sleep that includes both NREM and REM stages. The researchers will assess declarative memory performance, using a word-pair associates task, before and after the nap period for both the active and sham stimulation conditions. Autonomic physiology, including electrocardiography and impedance cardiography, will be gathered at baseline before the word-pairs task and continuously during sleep to examine vagal tone (i.e. heart rate variability) and sympathetic activation (i.e. pre-ejection period) in response to both the active and sham stimulation conditions. Polysomnography will also be gathered during the nap to examine sleep architecture.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult volunteers between the ages of 18-64.
* English speaking
* Self-reported napping

Exclusion Criteria:

* Aged greater than 64 years
* Lack of adherence to sleep/wake schedule of at least 7 hours a night for 5-days prior to study and during study timeline.
* Body mass index of 35 or above
* Presence of any clinical sleep disorder, including insomnia and obstructive sleep apnea (OSA)
* Presence of medical or psychiatric condition that is likely to affect sleep/wake function or cardiovascular functioning, including doctor diagnosed arrhythmia, bradycardia, hypertension, congestive heart failure, major depression, bipolar disorder, post-traumatic stress disorder.
* Medication use that is likely to affect sleep/wake function or cardiovascular functioning, including antidepressants, anxiolytic or soporific medication, and beta-blockers.
* Pregnancy
* Epilepsy
* head trauma
* alcoholism
* migraines
* metal pieces in the body (may confound tVNS delivery)
* history of substance abuse

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in memory between sham and active stimulation | active stimulation - sham stimulation (visits are counterbalanced); measured on day 6 and on day 12
  word-pair associates

SECONDARY OUTCOMES:
Change in amount of time in sleep stages between sham and active stimulation | active stimulation - sham stimulation (visits are counterbalanced); measured on day 6 and on day 12
  polysomnographically-recorded nap
Change in sleep spectral features between sham and active stimulation | active stimulation - sham stimulation (visits are counterbalanced); measured on day 6 and on day 12
  polysomnographically-recorded nap
Change in vagal activity between sham and active stimulation | active stimulation - sham stimulation (visits are counterbalanced); measured on day 6 and on day 12
  continuous heart rate variability during nap
Change in sympathetic activity between sham and active stimulation | active stimulation - sham stimulation (visits are counterbalanced); measured on day 6 and on day 12
  continuous impedance cardiography during nap

CONTACTS AND LOCATIONS:
Overall Officials: Lauren N Whitehurst, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Langley Porter Psychiatric Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark KB, Naritoku DK, Smith DC, Browning RA, Jensen RA. Enhanced recognition memory following vagus nerve stimulation in human subjects. Nat Neurosci. 1999 Jan;2(1):94-8. doi: 10.1038/4600. PMID 10195186
- [Background] Whitehurst LN, Cellini N, McDevitt EA, Duggan KA, Mednick SC. Autonomic activity during sleep predicts memory consolidation in humans. Proc Natl Acad Sci U S A. 2016 Jun 28;113(26):7272-7. doi: 10.1073/pnas.1518202113. Epub 2016 Jun 13. PMID 27298366
- [Background] Whitehurst LN, Naji M, Mednick SC. Comparing the cardiac autonomic activity profile of daytime naps and nighttime sleep. Neurobiol Sleep Circadian Rhythms. 2018 Mar 15;5:52-57. doi: 10.1016/j.nbscr.2018.03.001. eCollection 2018 Jun. PMID 31236511
- [Background] Kreuzer PM, Landgrebe M, Husser O, Resch M, Schecklmann M, Geisreiter F, Poeppl TB, Prasser SJ, Hajak G, Langguth B. Transcutaneous vagus nerve stimulation: retrospective assessment of cardiac safety in a pilot study. Front Psychiatry. 2012 Aug 7;3:70. doi: 10.3389/fpsyt.2012.00070. eCollection 2012. PMID 22891061
- [Background] Diekelmann S, Born J. The memory function of sleep. Nat Rev Neurosci. 2010 Feb;11(2):114-26. doi: 10.1038/nrn2762. Epub 2010 Jan 4. PMID 20046194
- [Background] Ghacibeh GA, Shenker JI, Shenal B, Uthman BM, Heilman KM. The influence of vagus nerve stimulation on memory. Cogn Behav Neurol. 2006 Sep;19(3):119-22. doi: 10.1097/01.wnn.0000213908.34278.7d. PMID 16957488
- [Background] Cellini N, Whitehurst LN, McDevitt EA, Mednick SC. Heart rate variability during daytime naps in healthy adults: Autonomic profile and short-term reliability. Psychophysiology. 2016 Apr;53(4):473-81. doi: 10.1111/psyp.12595. Epub 2015 Dec 16. PMID 26669510
- [Background] Clancy JA, Mary DA, Witte KK, Greenwood JP, Deuchars SA, Deuchars J. Non-invasive vagus nerve stimulation in healthy humans reduces sympathetic nerve activity. Brain Stimul. 2014 Nov-Dec;7(6):871-7. doi: 10.1016/j.brs.2014.07.031. Epub 2014 Jul 16. PMID 25164906